CLINICAL TRIAL: NCT04353401
Title: Whole Genome Sequencing Analysis of of SARS-CoV-2 Positive Patients
Brief Title: WGS Analysis of COVID-19 Positive Patients
Status: Completed | Type: Observational
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: VP-01-01; CALYPSO (Other: Vanda Pharmaceuticals)
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Coronavirus Infection; COVID-19
Keywords: Covid-19; WGS; viral load; viral genome
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We aim to better understand the mode of action of COVID-19 in the context of its interaction with the host genome through whole-genome sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Ability and acceptance to provide written informed consent and fluent in English.
* Men or women between 18-100+ years, inclusive.
* Willing to comply with study procedures.
* SARS-CoV-2 positive test result as confirmed by a RT-PCR assay with a sputum or nasopharyngeal sample (either done prior to or at the screening visit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 positive patients
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Associations with severity and outcomes | 3 months
  Clinical associations with human and viral genetics

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Investigational Site, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No